CLINICAL TRIAL: NCT00909818
Title: Hypofractionated Versus Standard Fractionated Whole Breast Irradiation to Node-negative Breast Cancer Patients: a Randomized Phase III Trial, CIRRO (The Lundbeck Foundation Center for International Research in Radiation Oncology)
Brief Title: Hypofractionated Versus Standard Fractionated Whole Breast Irradiation to Node-negative Breast Cancer Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Danish Breast Cancer Cooperative Group (Other)
Collaborators: Danish Cancer Society (Other)
Responsible Party: Principal Investigator, Birgitte Offersen, M.D., ph.d., associate professor, Danish Breast Cancer Cooperative Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DBCG hypo protocol; CIRRO IP030209; The Danish Cancer Society
Record Dates: First submitted 2009-05-28; First posted 2009-05-29 (Estimated); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Breast Cancer; Carcinoma in Situ of the Breast
MeSH Terms: conditions — Breast Neoplasms; Breast Carcinoma In Situ | interventions — Radiation Dose Hypofractionation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- standard fractionated radiotherapy (Active Comparator): 50 Gy/25 fractions, 2.00 Gy/fraction, 5 fractions per week
  Interventions: Radiation: standard fractionated radiotherapy
- hypofractionated radiotherapy (Experimental): hypofractionated radiotherapy 40 Gy/15 fractions
  Interventions: Radiation: hypofractionated radiotherapy

INTERVENTIONS:
Radiation: standard fractionated radiotherapy — standard fractionated radiotherapy 50 Gy/25 fractions
  Arms: standard fractionated radiotherapy
Radiation: hypofractionated radiotherapy — hypofractionated radiotherapy 40 Gy/15 fractions
  Arms: hypofractionated radiotherapy

SUMMARY:
The purpose of this study is to investigate the difference in late radiation morbidity between hypofractionated and standard fractionated breast irradiation given to women operated with breast conservation for early breast cancer.

DETAILED DESCRIPTION:
The randomization is between 50 Gy/25 fractions, 2.0 Gy per fraction, 5 fractions weekly, and 40 Gy/15 fractions, 2.67 Gy per fraction, 5 fractions weekly. The primary endpoint is late radiation morbidity; secondly, we want to investigate the frequency of local recurrences, and try to establish a genetic risk profile for development of late radiation morbidity.

The hypothesis is that women operated with breast conserving strategy for early breast cancer can be offered moderately hypofractionated radiotherapy without developing more late radiation morbidity compared to standard fractionated radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* operated with breast conserving strategy for:

  1. invasive breast cancer, pT1-2, pN0-1mi, M0 OR
  2. carcinoma in situ of the breast

Exclusion Criteria:

* previous radiation of the breast/thorax
* breast implants
* pregnant/lactating
* comorbidity which may hinder the patient in completing the therapy and complete follow up for 10 years

Min Age: 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 976 (Estimated)
Dates: Start 2009-05-14 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Grade 2 or 3 fibrosis 3 years after radiotherapy | 3 years

SECONDARY OUTCOMES:
Any other late morbidity after adjuvant radiotherapy, genetic risk profile for late morbidity, recurrence/survival | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Lars Stenbygaard, MD, Study Chair — Aalborg University Hospital; Birgitte Offersen, MD, Ph.D, Study Chair — Aarhus University Hospital; Erik Jakobsen, MD, Study Chair — Vejle Hospital; Mette H Nielsen, MD, phd, Study Chair — Odense University Hospital; Birgitte Offersen, MD, phd, Principal Investigator — Aarhus University Hospital; Mechthild Krause, M.D., Prof, Study Chair — University Clinic Carl Gustav Carus Dresden; Andreas Schreiber, M.D., Ph.D., Study Chair — Praxis für Strahlentherapie am Klinikum Dresden-Friedrichstadt; Ingvil Mjaaland, M.D., Study Chair — Helse Stavanger HF, Sorlandet Sykehus HF; Unn-Miriam Kasti, M.D., Study Chair — Kristiansand Sykehus
Locations (1):
- The Danish Breast Cancer Cooperative Group, Copenhagen, Denmark

REFERENCES:
- [Derived] Offersen BV, Alsner J, Nielsen HM, Jakobsen EH, Nielsen MH, Krause M, Stenbygaard L, Mjaaland I, Schreiber A, Kasti UM, Overgaard J; Danish Breast Cancer Group Radiation Therapy Committee. Hypofractionated Versus Standard Fractionated Radiotherapy in Patients With Early Breast Cancer or Ductal Carcinoma In Situ in a Randomized Phase III Trial: The DBCG HYPO Trial. J Clin Oncol. 2020 Nov 1;38(31):3615-3625. doi: 10.1200/JCO.20.01363. Epub 2020 Sep 10. PMID 32910709